CLINICAL TRIAL: NCT00482105
Title: Early Diagnosis of Melanoma Using Expression Profiling and Non-Invasive Sampling of Skin Cells
Acronym: DermTech
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn per sponsor and Investigator
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 200614850-1
Record Dates: First submitted 2007-05-31; First posted 2007-06-04 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Melanoma
Keywords: melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): This research study proposes to use a non-invasive method to capture superficial cells on pigmented skin lesions that are suspected of being early melanomas. This non-invasive "biopsy" technology has been developed and patented by DermTech International. RNA in skin cells captured by this method will be profiled in order to diagnose the nature of the lesion (i.e. malignant melanoma or not). A successful outcome of this proposal would create a candidate non-invasive diagnostic assay based on a gene expression profile for identifying early stage melanomas
  Interventions: Other: EGIR Tape

INTERVENTIONS:
Other: EGIR Tape — Tape stripping is a non-invasive method that allows the recovery of cells
  Other Names: Tape stripping (EGIR™)

SUMMARY:
This study is divided into distinct sample collection and analysis phases. In the sample collection phase investigators will tape strip lesions that are designated for biopsy because they are suspected for melanoma. No biopsies will be taken solely in support of this study; rather patients that present lesions that are to be biopsied-in the context of the standard of care-will be enrolled in the study and will have that lesion(s) tape stripped before the biopsy procedure.

In the second phase of the study, tape strip samples will be extracted and RNA purified and expression profiled by DNA microarray. The gene expression data will be correlated with histopathology with the expectation that an expression classifier that distinguishes suspect lesions from melanoma can be defined. That classifier will be validated in future studies.

DETAILED DESCRIPTION:
This is a multi-center study, sponsored by Derm Tech (DTI) International.

Specific Aims of the study

This research study proposes to use a non-invasive method to capture superficial cells on pigmented skin lesions that are suspected of being early melanomas. This non-invasive "biopsy" technology has been developed and patented by DermTech International. RNA in skin cells captured by this method will be profiled in order to diagnose the nature of the lesion (i.e. malignant melanoma or not). A successful outcome of this proposal would create a candidate non-invasive diagnostic assay based on a gene expression profile for identifying early stage melanomas. This assay and more in particular the diagnostic gene expression profile are considered candidate because the profile would have to be validated (i.e. proven to be diagnostic) in larger clinical trials. Secondary outcomes could include tests for diagnosis and prognosis of a variety of pigmented skin lesions.

Specific Aim 1: To create a sample set of pigmented skin lesions. Each sample consisting of:

1. RNA recovered by tape stripping the superficial epidermis overlying the lesion (tape stripping will also be used to recover RNA from normal skin areas and benign nevi as controls).
2. A standard biopsy of the same lesion and accompanying histology and diagnosis. Biopsies would be taken after tape stripping and subjected to standard histopathologic analysis, which would provide a "gold standard" diagnosis. These diagnoses could then be correlated with the data generated in Specific

Aim 2.

This specific aim is composed of three individual aims:

1. Analysis of selected lesion RNA samples by DNA microarray.
2. Correlation of gene expression data with histopathology.
3. Creation of a candidate expression classifier for diagnosis of melanoma.

Tape stripping (commercialized as a method for RNA recovery as Epidermal Genetic Information Retrieval or EGIR™) is a non-invasive method that allows recovery of cells comprising and associated with the upper epidermis [4]. The feasibility of non-invasive sampling of human epidermis by sequential adhesive tape stripping was shown by Morhenn et al [4]. Their work showed that tape stripping of skin yielded sufficient RNA for analysis by ribonuclease protection assay to detect specific RNA species, including those known to be at low abundance.

4. Therapeutically removed tissue will be collected

Tape-stripping procedure will be performed before all biopsy procedures. The tape will be applied to the site and briskly rubbed with the blunt rounded end of a marker or plastic test tube in a circular motion. A minimum of 15 circular motions must be completed before the tape is removed. To accommodate the fact that many sites will be smaller than the diameter of the tape, care will be taken to apply the tape only to the lesion or control site and not to the surrounding normal epidermis. The border of the lesion will be demarcated on the tape with a surgical marker; when the tapes are processed for RNA extraction, the marking will allow removal of tape that did not contact the lesion (and that might harbor normal epidermis). A total of 4 tapes will be used to sample a site greater than or equal to 6 mm in diameter. Preliminary data obtained from DTI show that lesions less than 6 mm in diameter may require up to 8 tapes to recover RNA. Tape stripping will also be performed on one normal appearing skin area (preferably; upper back or mastoid process) as well as one benign nevus (if available) to use as a comparison. After sampling, the tapes will be stored at -20oC or below. The tapes will be shipped to DTI on dry ice, by express mail, for analysis.

Biopsy After the tape-stripping procedure is completed, the whole lesion will be surgically excised according to standard clinical practice. The biopsy is a standard of care procedure that would be conducted regardless of the research. All tissues removed are fixed in formalin and sent to a histopathology laboratory, where they are embedded in paraffin and sectioned for histopathological analysis. Pathology results will be collected for distinguishing diagnosis. The subject pathology reports will be identified with the assigned unique subject identifiers prior to use in the study to protect subject identity.

ELIGIBILITY:
Inclusion Criteria:

The subject will be eligible if he or she:

* Is at least 18 years of age;
* Has a pigmented lesion that is suspected of being a melanoma and requires surgical removal.

Exclusion Criteria:

The subject cannot participate in this study if he or she:

* Has used topical medications (corticosteroids, alpha-hydroxyacids, or retinoids) within 30 days of beginning the research study;
* Has generalized skin disorders not related to skin cancer such as psoriasis, photosensitivity disorder or eczema;
* Has allergy to tape or latex rubber.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
A successful outcome of this proposal would create a candidate non-invasive diagnostic assay based on a gene expression profile for identifying early stage melanomas. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Tong Liu, M.D. PhD, Principal Investigator — UC Davis
Locations (1):
- UC Davis Department of Dermatology, Sacramento, California, United States

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical